CLINICAL TRIAL: NCT00684164
Title: Safety and Efficacy of Conivaptan for the Correction of Euvolemic and Hypervolemic Hyponatremia in Critically Ill Neurological Patients
Brief Title: Safety and Efficacy of Conivaptan for the Correction of Hyponatremia in Neurological Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to complete a contract with the Sponsor
Sponsor: Columbia University (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Stephan A. Mayer, MD, Columbia University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAC6833
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Hyponatremia
Keywords: Euvolemic Hyponatremia; Hypervolemic Hyponatremia; Neurological injury
MeSH Terms: conditions — Hyponatremia; Trauma, Nervous System | interventions — conivaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subjects in the treatment group will receive standard medical treatment plus Conivaptan administered as a 20mg bolus over 30 min, and then as a 20mg infusion over 24 hours for up to 4 days - or until the study endpoint of sodium ≥135mEq/L is reached.
  Interventions: Drug: Conivaptan
- 2 (Placebo Comparator): Subjects in the placebo control group will receive an equivalent volume loading dose of D5 followed by an infusion of D5 in the same manner as the experimental group.
  Interventions: Other: D5

INTERVENTIONS:
Drug: Conivaptan — 20mg bolus over 30 min, and then as a 20mg infusion over 24 hours for up to 4 days
  Other Names: VAPRISOL
  Arms: 1
Other: D5 — Volume loading dose of D5 followed by an infusion of D5 over 24 hours for up to 4 days - or until the study endpoint of sodium ≥135mEq/L is reached.
  Arms: 2

SUMMARY:
Low sodium levels (hyponatremia) are a frequent occurrence in medically ill patients, and in particular those with neurological injury. Hyponatremia has been associated with worse outcome, problems with memory and concentration and impaired balance. Standard treatment for low sodium (salt) levels is to give the patient a salt containing solution thru a catheter (small flexible tube) in a vein in the arm or leg. One of the major complications of this treatment is excess body fluid which may cause heart problems or accumulation of fluid in the lungs and may require additional medications to remove extra water from the body.

FDA approval has recently been granted for a new drug - Conivaptan - for use in hyponatremic conditions. Conivaptan works by excreting free water from the body and thereby produce concurrent rise in serum sodium concentrations. Conivaptan has not been evaluated specifically in patients with brain injuries. The primary objective of this study is to demonstrate the safety and efficacy of intravenous Conivaptan for the treatment of hyponatremia in patients with brain injury. If effective, Conivaptan may represent a safe treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Acute neurological injury
* Euvolemia or hypervolemia (defined clinically by examination, recent I+Os, BUN/creatinine ratio and CVP [if available])
* Serum sodium less than or equal to 132 mEq/L (confirmed as hypoosmolar hyponatremia by a concurrent source: osmolality measurements [<280 mosoms/L] or by a preceding serum Na+ value <135 mEq/L0

Exclusion Criteria:

* Patients who have uncontrolled hypertension; significant orthostatic hypotension or supine systolic blood pressure less than 85 mm Hg;
* Uncontrolled arrhythmias;
* Untreated severe hypothyroidism, hyperthyroidism, or adrenal insufficiency;
* Estimated creatinine clearance less than 20 ml/min;
* Urinary outflow obstruction unless catheterized;
* Alanine aminotransferase (ALT) >3x ULN
* Aspartate aminotransferase (AST) >3x ULN
* Serum albumin of 1.5 g/dl or less;
* Prothrombin time greater than 22 sec or an international normalized ratio (INR) greater than 2.0 without anticoagulant therapy or 3.0 or more with therapy; a white blood cell count less than 3000/µl;
* HIV infection;
* Active hepatitis.
* Pregnant or nursing
* Participation in a clinical trial of an investigational drug or device within 30 days of screening
* Unable to obtain written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2009-11 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Mean change in serum sodium over the duration of treatment between the two treatment arms. | From beginning of treatment to return of sodium level to greater than or equal to 135 mEq/L, up to 4 days of treatment

SECONDARY OUTCOMES:
Percentage of patients requiring study drug discontinuation for any reason other than reaching the sodium endpoint, including those with too rapid a rise in serum sodium (>12 mEq rise over 24 hours) or an infusion site reaction | From the initiation of treatment to the end of treatment, up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A. Mayer, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States